**Document:** TDOC-0056448 **Version:** 1.0; CURRENT; Most-Recent; Effective

Status: Effective

#### **Short Title:**

# Statistical Analysis Plan CLE383-C007/NCT03888469

#### **Full Title:**

# Statistical Analysis Plan CLE383-C007

**Protocol Title:** Clinical Comparison of DDT2 Contact Lens and a Daily

Disposable Contact Lens – Study 1

**Project Number:** A01660

**Protocol TDOC Number:** TDOC-0056080

Author:

**Template Version:** Version 4.0, approved 16MAR2015

**Approvals:** See last page for electronic approvals

**Job Notes:** 

This is the original (Version 1.0) Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 1.0 of the study protocol.


Status: Effective

**Executive Summary:** 

Key Objectives:

The primary objective of this study is to demonstrate noninferiority in visual acuity (VA) at distance when wearing Daily Disposable T2 Contact Lenses (DDT2) compared to 1-Day ACUVUE<sup>®</sup> Moist Contact Lenses (Acuvue Moist or Moist).

Decision Criteria for Study Success:

Success of this study will be based on demonstration of noninferiority in distance VA with DDT2 when compared to Moist, using a margin of 0.05.

Printed By: Print Date:


Status: Effective

## **Table of Contents**

Effective Date: 02-Apr-2019

| Statistic | cal Analysis Plan CLE383-C007 | 1 |
|-----------|-----------------------------------------------------|----|
| Table of | Contents | 3 |
| List of T | Tables | 4 |
| | Figures | |
| 1 | Study Objectives and Design | |
| 1.1 | Study Objectives | |
| 1.1 | Study Description | |
| 1.3 | Randomization | |
| 1.4 | Masking | |
| 1.5 | Interim Analysis | |
| 2 | Analysis Sets | |
| 2.1 | Safety Analysis Set | 7 |
| 2.2 | Full Analysis Set | |
| 2.3 | Per Protocol Analysis Set | 7 |
| 3 | Subject Characteristics and Study Conduct Summaries | 7 |
| 4 | Effectiveness Analysis Strategy | 8 |
| 4.1 | Effectiveness Endpoints | 9 |
| 4.2 | Effectiveness Hypotheses | 10 |
| 4.3 | Statistical Methods for Effectiveness Analyses | 11 |
| 4.3.1 | Primary Effectiveness Analyses | 11 |
| 4.6 | Interim Analysis for Effectiveness | 15 |
| 5 | Safety Analysis Strategy | 16 |
| 5.1 | Safety Endpoints | 16 |
| 5.2 | Safety Hypotheses | 16 |
| 5.3 | Statistical Methods for Safety Analyses | 16 |
| 5.3.1 | Adverse Events | |
| 5.3.2 | Biomicroscopy Findings | 17 |

| | | Effective Date: 02-Apr-2019 RRENT; Most-Recent; Effective |
|---|---|---|
| 5.3.3 | Device Deficiencies | 18 |
| 6 | Analysis Strategy for Other Endpo | ints18 |
| 7 | Sample Size and Power Calculation | ns18 |
| 8 | References | 19 |
| 9 | Revision History | 19 |
| 10 | Appendix | 20 |
| | List of | Tables |
| Table 1-1 | Study Description Summary | |
| Table 10-1 | Overview of Study Plan | 20 |
| | List of | Figures |
| Figure 1–1 | Study Design | 6 |


Status: Effective

# 1 Study Objectives and Design

## 1.1 Study Objectives

#### PRIMARY OBJECTIVE

The primary objective is to demonstrate noninferiority in distance VA when wearing DDT2 compared to Moist.



# 1.2 Study Description

Key components of the study are summarized in Table 1-1.

**Table 1-1 Study Description Summary** 

| Study Design | Design Prospective, randomized, bilateral crossover, double-masked, |
|---|---|
| | controlled |
| Study Population | Volunteer subjects aged 18 or over who are spherical soft contact |
| | lens wearers (excluding current/previous Moist and DAILIES |
| | TOTAL1® (DT1) lens wearers), and for the last 3 months have |
| | worn their habitual lenses at least 5 days per week and at least 8 |
| | hours per day in daily wear modality. |
| | Target to complete: 82 |
| | Planned to enroll: ~92 |
| Number of Sites | ~5 |
| | (US) |
| Test Product | Daily Disposable T2 Contact Lenses (Verofilcon A) (DDT2) |
| Control Product | 1-Day ACUVUE® MOIST Contact Lenses (etafilcon A) |
| | (Acuvue Moist or Moist) |
| Duration of Treatment | Up to 20 days total duration |
| | • Test Product: 8 days (-1/+2 days) |


Status: Effective

| | Control Product: 8 days (-1/+2 days) |
|--------|------------------------------------------------------------------|
| Visits | Visit 1* – Screening/Baseline/Dispense§ Lens 1 |
| | Visit 2 − 1-Week Follow-up Lens 1 at EOD/Dispense§ Lens 2 [8 |
| | days (-1/+2 days) from Visit 1] |
| | Visit 3 – 1-Week Follow-up Lens 2/Exit [8 days (-1/+2 days) from |
| | Visit 2] |
| | *Randomization will occur at Visit 1 |
| | §Study contact lens wear will commence day after each dispense |

A study design schematic is depicted in Figure 1–1.

Figure 1–1 Study Design

Visit 1
Screening / Baseline /
Dispense Lens 1

Visit 2
Follow-up Lens 1,
1 Week, EOD Visit
Dispense Lens 2

Visit 3
Follow-up Lens 2,
1 Week EOD Visit / Exit

#### 1.3 Randomization

A member of the Randomization Programming group at Alcon who is not part of the study team will generate the randomized allocation schedule(s) for study lens sequence assignment. Randomization will be implemented in

Qualifying subjects will be randomized in a 1:1 manner to one of 2 lens sequences consisting of the test lens and control lens as described below. For each sequence, subjects wear 1<sup>st</sup> lens then crossover to 2<sup>nd</sup> lens.

Sequence 1 = DDT2/Moist

Sequence 2 = Moist/DDT2


Status: Effective

#### 1.4 Masking

This study is double-masked.

#### 1.5 Interim Analysis

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination

#### 2 Analysis Sets

#### 2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study, except for the lenses used at Visit 1 for the purpose of parameter optimization and fitting, as they are not intended for the assessment of safety. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

Subjects who are lost to follow-up and their exposure to dispensed study lenses is unknown will be included in the safety analysis data set. The visit date for Dispense (Lens 1 or Lens 2) plus the presumed minimum 1 day of washout will be used as the first exposure date for the respective Lens.

Adverse events occurring from the time of informed consent but prior to first exposure to study lenses will be summarized in subject listings.

# **2.2** Full Analysis Set

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study lenses evaluated in this study, except for the lenses used for optimization and fitting.

## 2.3 Per Protocol Analysis Set

The per protocol (PP) analysis set is a subset of FAS and excludes all data/subjects that have met any of the critical deviation or evaluability criteria identified in the Deviation and Evaluability Plan (DEP).

# 3 Subject Characteristics and Study Conduct Summaries

The following tables will be presented:


Status: Effective

- Subject Disposition by Lens Sequence
- Analysis Sets by Lens Sequence
- Analysis Sets by Lens
- Subject Accounting by Lens Sequence
- Demographics Characteristics by Lens Sequence
- Baseline Characteristics by Lens Sequence (eg, summary statistics for subjective ratings)

Demographic characteristics and subject accounting tables will be summarized by lens sequence and overall on the safety, full, and per protocol analysis datasets. Baseline characteristics will be summarized by lens sequence and overall on the full and per protocol analysis datasets.

In addition, the following subject listings will be provided:

- Listing of Subjects Excluded from Protocol Defined Analysis Sets
- Listing of Lens Sequence Assignment by Investigator
- Listing of Subjects Discontinued from Study

#### 4 Effectiveness Analysis Strategy

| This study defines one primary, |
|---------------------------------|
| FAS as the primary |

Continuous variables will be summarized using the number of observations, mean, standard deviation, median, minimum and maximum, as well as confidence intervals/limits as applicable. Categorical variables will be summarized with counts and percentages from each category.

| All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation |
|---|
| for missing values will be carried out |


Status: Effective



Effective Date: 02-Apr-2019

## 4.1 Effectiveness Endpoints

#### **Primary Endpoint**

The primary endpoint is VA at distance with study lenses, collected separately for each eye in logMAR.



Status: Effective



# 4.2 Effectiveness Hypotheses

## **Primary Effectiveness**

The null and alternative hypotheses for the primary analysis are formulated in terms of the predefined margin of 0.05 for noninferiority:

$$H_0$$
:  $\mu_{(T)}$  -  $\mu_{(C)} \! \geq \! 0.05$ 

$$H_a$$
:  $\mu_{(T)}$  -  $\mu_{(C)}$   $\!<$   $\!0.05$ 

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the mean distance VA for DDT2 and Moist, respectively, on the logMAR scale.




Effective Date: 02-Apr-2019


Status: Effective



# 4.3 Statistical Methods for Effectiveness Analyses

## 4.3.1 Primary Effectiveness Analyses

A mixed effects repeated measures model will be utilized to test these hypotheses. The model will include terms for lens, period, and sequence. Within-subject correlation due to eye and the crossover design will also be accounted for in the model. Lens difference (DDT2 minus Moist) and the corresponding one-sided 95% upper confidence limit will be computed. Noninferiority in distance VA will be declared if upper confidence limit is less than 0.05.



Printed By: Print Date:

Effective Date: 02-Apr-2019

Alcon - Business Use Only Statistical Analysis Plan Version: 1.0; CURRENT; Most-Recent; Effective Document: TDOC-0056448 Status: Effective

Printed By: Print Date: Effective Date: 02-Apr-2019

Effective Date: 02-Apr-2019 Version: 1.0; CURRENT; Most-Recent; Effective Document: TDOC-0056448

Status: Effective




Status: Effective



# 4.6 Interim Analysis for Effectiveness

No interim analysis is planned for the effectiveness endpoints.

Printed By: Print Date:

Effective Date: 02-Apr-2019


Status: Effective

#### 5 Safety Analysis Strategy

## 5.1 Safety Endpoints

The safety endpoints are:

- Adverse events (AE)
- Biomicroscopy findings
  - Limbal hyperemia (also an exploratory effectiveness endpoint)
  - Bulbar hyperemia (also an exploratory effectiveness endpoint)
  - Corneal staining
  - Conjunctival staining
  - o Palpebral conjunctival observations
  - Corneal epithelial edema
  - Corneal stromal edema
  - o Corneal vascularization
  - Conjunctival compression/indention
  - o Chemosis
  - o Corneal infiltrates
  - Other findings
- Device deficiencies

## 5.2 Safety Hypotheses

There are no formal safety hypotheses in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.

# 5.3 Statistical Methods for Safety Analyses

The analysis set for all safety analyses is defined in Section 2.1. Baseline will be defined as the last measurement prior to exposure to study lenses. For biomicroscopy data, baseline will be defined as Visit 1 for Period 1 and Visit 2 for Period 2. Safety variables will be summarized descriptively.

#### 5.3.1 Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs informed consent to when a subject exits the study will be accounted for in the reporting.


Status: Effective

Analysis and presentation of pre-treatment AEs and between-treatment AEs will be separated from treatment-emergent AEs occurring during the study periods. A pre-treatment AE is an event that occurs after signing informed consent but prior to exposure to study lenses. A between-treatment AE is an event that occurs after last exposure to Period 1 lenses but prior exposure to Period 2 lenses. The period for treatment-emergent AE analysis starts from exposure to study lenses for Period 1 or Period 2 until the subject completes the respective period or is discontinued from the study.

The following tables and supportive listings will be provided:

- Incidence of All Ocular Treatment-Emergent Adverse Events
- Incidence of Ocular Serious Treatment-Emergent Adverse Events
- Incidence of Ocular Significant Non-serious Treatment-Emergent Adverse Events
- Incidence of All Nonocular Treatment-Emergent Adverse Events
- Incidence of Nonocular Serious Treatment-Emergent Adverse Events
- Listing of All Ocular Treatment-Emergent Adverse Events
- Listing of All Nonocular Treatment-Emergent Adverse Events
- Listing of All Ocular Pre-Treatment Adverse Events
- Listing of All Nonocular Pre-Treatment Adverse Events
- Listing of All Ocular Between-Treatment Adverse Events
- Listing of All Nonocular Between-Treatment Adverse Events

## 5.3.2 Biomicroscopy Findings

The following tables and supportive listings will be provided:

- Frequency and Percentage for Biomicroscopy Findings by Visit
- Incidence of Increased Severity by 2 or More Grades in Biomicroscopy Findings
- Listing of Subjects With Other Biomicroscopy Findings
- Listing of Subjects With Increased Severity by 1 Grade in Biomicroscopy Findings [This listing will include all relevant visits within the crossover period]
- Listing of Subjects With Increased Severity by 2 or More Grades in Biomicroscopy Findings [This listing will include all relevant visits within the crossover period]
- Listings of Subjects with Infiltrates


Status: Effective

#### **5.3.3** Device Deficiencies

The following tables and supportive listings will be provided:

- Frequency of Treatment-Emergent Device Deficiencies
- Listing of Treatment-Emergent Device Deficiencies
- Listing of Device Deficiencies Prior To Treatment Exposure

#### 6 Analysis Strategy for Other Endpoints

Not applicable

## 7 Sample Size and Power Calculations

Sample size calculation is based on a prior clinical study (CLE383-C004) which evaluated performance of DDT2 and 3 marketed soft contact lenses, including Acuvue Moist.

#### **Primary Effectiveness**

To demonstrate noninferiority (margin = 0.05 in logMAR;  $\frac{1}{2}$  line in Snellen) in distance VA as a one-tailed hypothesis with  $\alpha$ =0.05, and using a standard deviation of 0.068 for paired differences, 80% power can be attained with a sample size of 14 (7 per sequence).




Status: Effective

# **8** References

# 9 Revision History

This is the original (Version 1.0) Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 1.0 of the study protocol.

Alcon - Business Use Only Statistical Analysis Plan
Status: Effective

#### Appendix **10**

**Table 10-1** Overview of Study Plan

| Procedure / Assessment | Visit 1 Screening / Baseline / Dispense Lens 1 (Lens 1 to be worn after washout period) | Visit 2<br>1-Week Follow-up<br>Lens 1 at EOD□ /<br>Dispense Lens 2 | Visit 3<br>1-Week Follow-up<br>Lens 2 at EOD□ / Exit | Unscheduled Visit /<br>Early Exit |
|---|---|---|---|---|
| | Washout period: Subjects will<br>discontinue habitual lens wear<br>after the screening visit until<br>the next day when they<br>commence wearing study<br>Lens 1∞ | 8 (-1/+2) days after Visit 1 Washout period: Subjects will wear spectacles after Visit 2 until the next day when they commence wearing study Lens 2.∞ | 8 (-1/+2) days after Visit 2 | N/A |
| Informed Consent | ✓ | - | - | - |
| Demographics | ✓ | - | - | - |
| Medical History | ✓ | ✓ | ✓ | ✓ |
| Concomitant Medications | ✓ | ✓ | ✓ | ✓ |
| Inclusion / Exclusion | ✓ | - | - | - |
| Habitual lens information (brand, power)* | ✓ | - | - | - |
| VA with habitual contact lens correction (OD, OS, Snellen distance)* | ✓ | - | ✓ (Exit procedure) | (✔) |
| | ✓ | - | - | - |
| BCVA (Snellen distance with manifest refraction) OD, OS* | ✓ | (✔) | (✔) | (✔) |
| Biomicroscopy | ✓ | ✓ | ✓ | ✓ |
| Fit both study products (lenses) using fitting guide | ✓ | - | - | - |
| | | - | - | - |
| Dispense (provide) study lenses | ✓ | ✓ | - | (✓) |
| VA (logMAR distance) with study lenses, OD, OS | ✓* (with both fitting set lens types) | ✓ | ✓ | (✓) |

Alcon - Business Use Only Statistical Analysis Plan
Status: Effective

| Procedure / Assessment | Visit 1 Screening / Baseline / Dispense Lens 1 (Lens 1 to be worn after washout period) | Visit 2<br>1-Week Follow-up<br>Lens 1 at EOD□ /<br>Dispense Lens 2 | Visit 3<br>1-Week Follow-up<br>Lens 2 at EOD□ / Exit | Unscheduled Visit /<br>Early Exit |
|---|---|---|---|---|
| | Washout period: Subjects will<br>discontinue habitual lens wear<br>after the screening visit until<br>the next day when they<br>commence wearing study<br>Lens 1∞ | 8 (-1/+2) days after Visit 1 Washout period: Subjects will wear spectacles after Visit 2 until the next day when they commence wearing study Lens 2.∞ | 8 (-1/+2) days after Visit 2 | N/A |
| | | | | - |
| | I | <b>=</b> | | I |
| AEs | ✓ | ✓ | ✓ | ✓ |
| Device Deficiencies | ✓ | ✓ | ✓ | ✓ |
| Exit Form | (✓) | (✓) | (✓) | (✓) |
| * source only | (✓) assessment performed | as necessary, eg, decrease | of VA by 2 lines or more w | ith investigational product |


Status: Effective


Effective Date: 02-Apr-2019

Status: Effective

| Signed by: | Justification: |
|------------|----------------|